CLINICAL TRIAL: NCT01158183
Title: Real-World Betaseron® Outcomes Study (ROBUST): A Twelve-month, US Prospective, Observational, Open-label, Single-arm, Multi-center Outcomes Study of Interferon β-1b (Betaseron®) Given Every Other Day for Relapsing Forms of Multiple Sclerosis
Brief Title: Real-World Betaseron Health Economic Outcomes Study for Relapsing Forms of Multiple Sclerosis
Acronym: ROBUST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare Pharmaceuticals Inc.
Other Study IDs: 14838; BF0714US; 311644
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Outcomes; real world and web tool; electronic data capture
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: No intervention
  Interventions: Drug: BAY86-5046_Interferon-beta-1b

INTERVENTIONS:
Drug: BAY86-5046_Interferon-beta-1b — Electronic questionnaires

SUMMARY:
A Web based real world observational study in Relapsing-Remitting Multiple Sclerosis (RRMS) population capturing outcomes reported by patients and by the physicians during 12 months after initiating or resuming Betaseron.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent to participate in the study
* At least 18 but no more than 65 years old
* Documented clinical diagnosis of a relapsing form of multiple sclerosis or confirmed clinically isolated syndrome (CIS)
* Initiating Betaseron therapy, or resuming Betaseron after not having used it for at least three months
* Willing and able to provide a valid e-mail address which will be in use for the duration of the study
* Willing and able to complete study questionnaires via the Internet
* Has reliable Internet access for the duration of the study
* Completes the baseline patient questionnaire

Exclusion Criteria:

* Kurtzke Expanded Disability Status Scale (EDSS) score greater than 6.0
* Cognitive dysfunction that, in the Investigator's judgment, raises doubts about the study participant's ability to provide informed consent or accurately complete the monthly patient questionnaire
* Any use of Betaseron within the three months prior to study entry
* Inability to read, write, or speak the English language
* Illness or disease other than multiple sclerosis that the Investigator believes is likely to cause the patient's death or incapacity within twelve months
* Any severe, uncontrolled illness or condition that the Investigator believes could dominate the patient's quality of life
* Coexistent autoimmune disease such as rheumatoid arthritis, lupus, or psoriasis that is likely to be exacerbated by treatment with Interferon
* Current use of any immunosuppressive medication
* Previous participation in a multiple sclerosis (MS) clinical trial within the three months prior to study entry
* Previous use of monoclonal antibodies treating MS within the three months prior to study entry
* Current use of any secondary treatment for multiple sclerosis other than the episodic use of steroids during relapses or exacerbations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "real world" population
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Key Objective: To collect patient reported outcomes and clinical assessments via the same web-based data capture tool in a real world setting in relapse-remitting multiple sclerosis patients | Baseline, 1 to12 month outcome questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- United States (27):
  - Many Locations, Alabama
  - Many Locations, California
  - Many Locations, Colorado
  - Many Locations, Florida
  - Many Locations, Illinois
  - Many Locations, Iowa
  - Many Locations, Kansas
  - Many Locations, Louisiana
  - Many Locations, Maine
  - Many Locations, Massachusetts
  - Many Locations, Michigan
  - Many Locations, Missouri
  - Many Locations, Nevada
  - Many Locations, New Hampshire
  - Many Locations, New Jersey
  - Many Locations, New York
  - Many Locations, North Carolina
  - Many Locations, North Dakota
  - Many Locations, Ohio
  - Many Locations, Oregon
  - Many Locations, Pennsylvania
  - Many Locations, Rhode Island
  - Many Locations, Tennessee
  - Many Locations, Texas
  - Many Locations, Virginia
  - Many Locations, Washington
  - Many Locations, Wisconsin